CLINICAL TRIAL: NCT01749761
Title: Blood Pressure Guided Biofeedback on Hemodialysis and the Reduction of IntraDialytic Hypotensive Episodes: A Randomized Cross Over Trial
Brief Title: Blood Pressure Guided Biofeedback on Hemodialysis and the Reduction of IntraDialytic Hypotension
Acronym: BP-RIDH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of British Columbia (Other); B. Braun Medical Inc. (Industry)
Responsible Party: Principal Investigator, Dr Jennifer MacRae, Primary Investigator, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H12-02619
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Hypotension
Keywords: IDH, intradialytic hypotension,; hypotension on hemodialysis,; hemodialysis,; Blood pressure guided biofeedback
MeSH Terms: conditions — Hypotension | interventions — Renal Dialysis; Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemodialysis without biofeedback (Placebo Comparator): Patients will be randomized to receive hemodialysis without biofeedback for a period of 8 weeks.
  Interventions: Other: BioLogic RR
- BioLogic RR biofeedback (Active Comparator): Patients will receive 8 weeks of HD with BioLogic RR Blood pressure guided biofeedback.
  Interventions: Other: Hemodialysis without biofeedback

INTERVENTIONS:
Other: BioLogic RR — Patients will be randomized to BP guided biofeedback arm which will entail regular hemodialysis with a software program turned on to allow frequent assessment of blood pressure and automated adjustments of the ultrafiltration rate based on these blood pressure measurements. The duration of this arm is 8 weeks
  Other Names: BioLogics Comfort RR, B Braun software
  Arms: Hemodialysis without biofeedback
Other: Hemodialysis without biofeedback — patients will be randomized to Standard HD (without biofeedback technology) for 8 weeks
  Other Names: Hemodialysis
  Arms: BioLogic RR biofeedback

SUMMARY:
It is very common for hemodialysis patients to have problems with low blood pressure while on hemodialysis. Low blood pressure on dialysis is not a good thing and it is associated with an increased risk of death and hospitalizations. It might be possible to minimize or even prevent these low blood pressure episodes with a software that can be added to the dialysis machine which detects the patient's changes in blood pressure and automatically slows down how much fluid is being removed from the person.

The investigators hypothesize that a blood pressure guided biofeedback system (called BioLogics RR) will result in a 30% reduction in the number of hypotensive episodes on hemodialysis.

DETAILED DESCRIPTION:
This is a randomized cross over trial in which 30 chronic hemodialysis patients with a history of intradialytic hypotension, IDH will be randomized to receive either standard hemodialysis or hemodialysis with blood pressure guided biofeedback (BioLogics RR Comfort, B braun). After the initial period of 8 weeks patients will cross over to the other group for the final 8 weeks of the study.

The primary outcome is the reduction in the number of IDH episodes associated with patient symptoms or nursing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* chronic hemodialysis patients
* history of 3 of the last 12 runs with documented hypotension with symptoms or nursing interventions

Exclusion Criteria:

* <19 years
* hemodiafiltration
* expected switch in modality within next 6 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
intradialytic hypotension episodes | By the end of the 8 week intervention period
  A 30% reduction in the frequency of HD sessions complicated by IDH. IDH is defined as a reduction in systolic BP of > = 20 mmHg if the pre-dialysis BP is >= 100 mmHg and with patient symptoms or nursing intervention. IDH is defined as a reduction in systolic BP of >=10 mmHg if predialysis BP < = 90mm Hg and with patient symptoms or nursing interventions

SECONDARY OUTCOMES:
urea clearance | 8 weeks
  Change in urea clearance
Brain natriuretic peptide | 8 weeks
  change in BNP
intradialytic hypotension (blood pressure criteria alone) | 8 weeks
  Reduction in the number of IDH episodes based on BP criteria alone
Intradialytic symptoms | 8 weeks
  Reduction in the number of intradialytic symptoms

OTHER OUTCOMES:
Oxygenation saturation | 8 weeks
  Reduction in the minimum 02 saturation achieved

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M MacRae, MD, Principal Investigator — University of Calgary
Locations (1):
- St.Paul's Hospital Hemodialysis Unit, Vancouver, British Columbia, Canada